CLINICAL TRIAL: NCT05236920
Title: Utility and Procedural Feasibility of REBOA Operationalized for Non-Trauma Application (UP-FRONT)
Acronym: UP-FRONT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study will not take place at this time.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Michael C. Kurz, Professor and Vice Chair for Research, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300007924
Record Dates: First submitted 2022-01-14; First posted 2022-02-11 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Ventricular Fibrillation; Ventricular Tachycardia
Keywords: cardiac arrest; out of hospital cardiac arrest; REBOA
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation; Tachycardia, Ventricular; Heart Arrest

STUDY DESIGN:
Intervention Model Description: A total of 40 subjects will be randomized to standard care, or standard care plus administration of the device.
Masking Description: None. Masking is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Care (No Intervention): Participants randomized to this arm will receive standard care for cardiac arrest, which consists of advanced cardiovascular life support (ACLS)
- Standard Care Plus Intervention (Experimental): Participants randomized to this arm will receive standard care for cardiac arrest, which consists of advanced cardiovascular life support (ACLS) plus the study intervention
  Interventions: Device: Resuscitative Endovascular balloon occlusion of the aorta using a REBOA catheter device

INTERVENTIONS:
Device: Resuscitative Endovascular balloon occlusion of the aorta using a REBOA catheter device — In-hospital use of a REBOA catheter device during advanced cardiac life support
  Other Names: REBOA procedure
  Arms: Standard Care Plus Intervention

SUMMARY:
Single center randomized-controlled trial in out-of-hospital cardiac arrest (OHCA) patients. This study will investigate the feasibility and utility of the Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) procedure using a REBOA catheter device in patients who have experienced an OHCA and have not regained return of spontaneous circulation (ROSC).

DETAILED DESCRIPTION:
Victims arriving to, or experiencing witnessed Ventricular Fibrillation (VF) or Ventricular Tachycardia (VT) out of hospital cardiac arrest in, the UAB emergency department with greater than 10 minutes of conventional ACLS will be eligible. The study population will consist of forty (40) subjects randomized to either continued contemporary standard of care (ACLS), or ACLS plus the administration of a REBOA catheter device.

The aims of UPFRONT are:

1. To describe the feasibility of rapid deployment of a REBOA catheter device in the setting of OHCA
2. To evaluate the utility of a REBOA catheter device to achieve ROSC in the setting of OHCA.

ELIGIBILITY:
Inclusion Criteria:

1. Apparent age between 18 - 70 years.
2. OHCA defined as receiving professional CPR or AED defibrillation
3. OHCA witnessed by bystanders or professional rescuers / UED personnel
4. VT/VF as the presenting rhythm for OHCA or clearly documented VT/VF during OHCA
5. Total time pulseless > 10 minutes

Exclusion Criteria:

1. Obvious Pre-existing neurocognitive impairment precluding independent activities of daily living
2. Obvious or suspicion of anatomic abnormality preventing successful deployment of REBOA device (i.e. previous vascular surgery in access region, dialysis graft, etc.)
3. Clear non-cardiac etiology (traumatic, hanging, overdose, etc.) of cardiac arrest
4. Do-Not-Resuscitate order or comfort care measures in place prior to enrollment
5. Special populations (pregnant, prisoner, or cognitively impaired)
6. Total time pulseless greater than 20 minutes
7. Inability to determine when cardiac arrest occurred (or for OHCA arriving to UED via EMS, time of 911 call) and the time elapsed since

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Time to successful deployment of device | Up to 10 minutes
  The device is successfully deployed when it raises the mean arterial pressure

SECONDARY OUTCOMES:
Return of spontaneous circulation (ROSC) | Up to 60 minutes
  ROSC is when the heart begins beating on its own

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Kurz, MD, Principal Investigator — Professor and Vice-Chair for Research, Department of Emergency Medicine

IPD SHARING:
Plan to Share IPD: No
The investigator has no plans to share individual participant data with other researchers. Any future use of the data will be proposed to and approved by the Principal Investigator, and will require IRB approval.